CLINICAL TRIAL: NCT03175289
Title: The Impact of Expiratory Muscle Strength Training on Bulbar Function and Well Being of Individuals With Head and Neck Cancer
Brief Title: Expiratory Muscle Strength Training in Improving Bulbar Function and Quality of Life in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16023; NCI-2017-00848 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care, home exercises) (Active Comparator): Patients receive standard of care comprising of written patient education materials focusing on oral care, signs/symptoms of dysphagia/aspiration, and trismus. Patients participate in a therapy session conducted by a speech pathologist over 30 minutes once per week for 6 weeks during chemoradiation therapy. Patients also perform prescribed exercises at home daily for 3 sets of 10 repetitions.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard of care, home exercises, EMST) (Experimental): Patients receive standard of care comprising of written patient education materials focusing on oral care, signs/symptoms of dysphagia/aspiration, and trismus. Patients participate in a therapy session conducted by a speech pathologist over 30 minutes once per week for 6 weeks during chemoradiation therapy. Patients perform prescribed exercises at home daily for 3 sets of 10 repetitions. Patients also participate in an EMST session over 30 minutes comprising of 5 sets of 5 repetitions daily for 5 days per week for 6 weeks during chemoradiation therapy
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Exercise Intervention; Other: Expiratory Muscle Strength Training; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo therapy session conducted by a speech pathologist
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive standard of care patient education materials focusing on oral care, signs/symptoms of dysphagia/aspiration, and trismus
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Exercise Intervention — Perform prescribed home exercises
Other: Expiratory Muscle Strength Training — Participate in EMST
  Other Names: EMST
  Arms: Arm II (standard of care, home exercises, EMST)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well expiratory muscle strength training works in improving bulbar function and quality of life in patients with head and neck cancer. Expiratory muscle strength training may help to strengthen the muscles involved in breathing and swallowing and may allow improved breathing, airway safety, swallow function, and quality of life in patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Investigate the impact of a prophylactic targeted exercise program, expiratory muscle strength training (EMST), on swallowing function and well-being of individuals on head and neck cancer (HNC).

II. Determine the impact of EMST on objective respiratory measures of individuals with HNC.

III. Determine the relationship between mean dose across the swallowing muscles (oral tongue and supra-hyoids, base of tongue, superior, middle and inferior pharyngeal constrictors, proximal esophagus)/dose on each muscle and the swallowing functional outcomes from aim 1.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care comprising of written patient education materials focusing on oral care, signs/symptoms of dysphagia/aspiration, and trismus. Patients participate in a therapy session conducted by a speech pathologist over 30 minutes once per week for 6 weeks during chemoradiation therapy. Patients also perform prescribed exercises at home daily for 3 sets of 10 repetitions.

ARM II: Patients receive standard of care comprising of written patient education materials focusing on oral care, signs/symptoms of dysphagia/aspiration, and trismus. Patients participate in a therapy session conducted by a speech pathologist over 30 minutes once per week for 6 weeks during chemoradiation therapy. Patients perform prescribed exercises at home daily for 3 sets of 10 repetitions. Patients also participate in an EMST session over 30 minutes comprising of 5 sets of 5 repetitions daily for 5 days per week for 6 weeks during chemoradiation therapy.

After completion of study, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definitive, curative treatment plan consisting of chemoradiation for head & neck cancer

  * Surgery, if required, must be limited to: diagnostic biopsy

Exclusion Criteria:

* Participants enrolled in a radiation de-intensification protocol
* Current or previous neurological disease, which may adversely affect swallowing
* History of oropharyngeal swallowing disorder prior to cancer diagnosis
* Previous neurosurgery on the brain
* Severe chronic obstructive pulmonary disease (COPD) requiring oxygen dependence, as this is a contraindication of EMST

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Airway safety during swallowing assessed using the Penetration-Aspiration Scale | Up to 1 year
  Exploratory mixed effect model will be used to investigate swallow function with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.

SECONDARY OUTCOMES:
Eating Assessment Tool-10 | Up to 1 year
  Collected variables will be estimated through patient and clinician surveys.
Expiratory flow assessed using portable digital peak flow meter | Up to 1 year
  Exploratory mixed effect model will be used to investigate respiratory measures with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.
Functional Oral Intake Scale (FOIS) | Up to 1 year
  Collected variables will be estimated through patient and clinician surveys.
Lingual strength defined as the maximum pressure of the tongue pressing against the hard palate measured using the Iowa Oral Performance Instrument | Up to 1 year
  Exploratory mixed effect model will be used to investigate swallow function with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.
Maximum expiratory pressure assessed using the MicroRPM pressure meter | Up to 1 year
  Exploratory mixed effect model will be used to investigate respiratory measures with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.
Maximum mandibular opening using the TheraBite range of motion scale | Up to 1 year
  Exploratory mixed effect model will be used to investigate swallow function with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.
Patient reported quality of life assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | Up to 1 year
  Exploratory mixed effect model will be used to investigate quality of life with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable.
Respiratory-swallow phase patterns captured using the standard Modified Barium Swallow Study | Up to 1 year
  Logistic regression method will be used to explore associations between treatment and respiratory-swallow phase (normal/abnormal).
Swallow pathophysiology assessed using the Modified Barium Swallow Impairment Profile | Up to 1 year
  Exploratory mixed effect model will be used to investigate swallow function with time (pre and 1, 3, 6, and 12 month post) as the within-subjects variable and group (expiratory muscle strength training and control) as the between-subjects variable. Pearson or Spearman correlation methods will be used to evaluate the relationship between swallow function/patterning and respiratory and swallow safety measures.

CONTACTS AND LOCATIONS:
Overall Officials: Loni Arrese, PhD, SLP, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu